CLINICAL TRIAL: NCT06490536
Title: A Precision Medicine Trial Leveraging Blood-Based Tumor Genomics to Optimize Treatment in Operable Stage III and High-Risk Stage II Colon Cancer Patients
Brief Title: The Sagittarius Trial
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: IFOM ETS - The AIRC Institute of Molecular Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IFOM-CPT009/2022/PO008; 2023-509851-15-00 (EU CTIS Number)
Record Dates: First submitted 2024-06-11; First posted 2024-07-08 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Colon Cancer Stage II; Colon Cancer Stage III
MeSH Terms: conditions — Colonic Neoplasms | interventions — Oxaliplatin; Capecitabine; Leucovorin; Fluorouracil; Temozolomide; Irinotecan; Nivolumab; Ipilimumab; Trastuzumab; pertuzumab; Panitumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (6):
- Trial-1 (ctDNA+) Strata-1 (MSS/MMRp extendend RAS/RAFmut) Standard Therapy (Active Comparator): CAPOX/FOLFOX for 6 months or until toxicity
  Interventions: Drug: Oxaliplatin; Drug: Capecitabine; Drug: Folinic acid; Drug: Fluorouracil
- Trial-1 (ctDNA+) Strata-1 (MSS/MMRp extendend RAS/RAFmut) Tailored Therapy (Experimental): CAPOX for 3 months with an interventional liquid biopsy at the end of the treatment. Patients still resulting ctDNA+ will be switched to a tailored therapy (FOLFIRI for RAS/RAF-mutated and MGMT-positive tumors or TEMIRI for RAS/RAF-mutated and MGMT-negative tumors) for 6 months or until toxicity. On the other hand, ctDNA- patients will continue CAPOX up to 3 months, and their ctDNA status will be re-assessed at the end of the treatment. Patients remaining ctDNA- will enter into follow-up, while patients resulting ctDNA+ will be switched to the tailored therapy.
  Interventions: Drug: Oxaliplatin; Drug: Capecitabine; Drug: Folinic acid; Drug: Fluorouracil; Drug: Temozolomide; Drug: Irinotecan
- Trial-1 (ctDNA+) Strata-2 (MSI-H/MMRd & MSS/MMRp extended RAS/RAFwt) Standard Therapy (Active Comparator): CAPOX/FOLFOX for 6 months or until toxicity
  Interventions: Drug: Oxaliplatin; Drug: Capecitabine; Drug: Folinic acid; Drug: Fluorouracil
- Trial-1 (ctDNA+) Strata-2 (MSI-H/MMRd & MSS/MMRp extended RAS/RAFwt) Tailored Therapy (Experimental): Tailored therapy (nivolumab+ipilimumab for MSI-H/MMRd: MSI-H/MMRd tumors and MSS/MMRp tumors with POLE mutations and a high TMB or trastuzumab + pertuzumab for MSS/MMRp HER2-amplified tumors or panitumumab+folfox for MSS/MMRp RAS/RAF/HER2 wild-type) for 3 months, at the end, the ctDNA status of patients will be reassessed to further guide their subsequent treatments. Patients still ctDNA+ at will be switched to standard therapy. On the other hand, patients undergoing seroconversion will continue the same therapy for 3 further months and will be then re-assessed at the end of the treatment. Patients resulting ctDNA- will enter into Follow-up, while patients resulting ctDNA+ will be switched to the standard therapy.
  Interventions: Drug: Nivolumab; Drug: Ipilimumab; Drug: Trastuzumab; Drug: Pertuzumab; Drug: Panitumumab
- Trial-2 (ctDNA-) Standard Therapy (Active Comparator): Chemotherapy regimen at prior declared physician choice (CAPE/CAPOX/FOLFOX/5-FU±LV).
  Interventions: Drug: Oxaliplatin; Drug: Capecitabine; Drug: Folinic acid; Drug: Fluorouracil
- Trial-2 (ctDNA-) Intensive Follow-up (No Intervention): Intensive follow-up for 6 months (except for MSS Stage III High-risk patients which will be treated with CAPE).

INTERVENTIONS:
Drug: Oxaliplatin — Oxaliplatin is used as part of the chemotherapy regimens for patients with ctDNA+ results in the SAGITTARIUS trial. It is administered in the following ways:
  CAPOX Regimen: Oxaliplatin 130 mg/m² is given intravenously on day 1, in combination with capecitabine 1000 mg/m² taken orally twice daily on days 1-14 of each 21-day cycle.
  FOLFOX Regimen: Oxaliplatin 85 mg/m² is administered intravenously on day 1, alongside folinic acid 400 mg/m² and fluorouracil 400 mg/m² IV bolus, followed by 2400 mg/m² IV infusion over 46 hours, in each 14-day cycle.
  Dosages are standardized, while the duration of treatment can be adjusted based on patient response and liquid biopsy results, typically up to 6 months.
  Arms: Trial-1 (ctDNA+) Strata-1 (MSS/MMRp extendend RAS/RAFmut) Standard Therapy; Trial-1 (ctDNA+) Strata-1 (MSS/MMRp extendend RAS/RAFmut) Tailored Therapy; Trial-1 (ctDNA+) Strata-2 (MSI-H/MMRd & MSS/MMRp extended RAS/RAFwt) Standard Therapy; Trial-2 (ctDNA-) Standard Therapy
Drug: Capecitabine — Capecitabine is used as part of the chemotherapy regimens for patients with ctDNA+ and ctDNA- results in the SAGITTARIUS trial. It is administered in the following ways:
  CAPOX Regimen: Capecitabine 1000 mg/m² is taken orally twice daily on days 1-14 of each 21-day cycle, in combination with oxaliplatin 130 mg/m² given intravenously on day 1.
  Capecitabine Monotherapy for High-Risk ctDNA- Patients: Capecitabine 1250 mg/m² is taken orally twice daily on days 1-14 of each 21-day cycle for patients identified as high-risk but with negative ctDNA results.
  The dosage of capecitabine is standardized, while the duration of treatment varies based on patient response and monitoring results, typically up to 6 months.
  Arms: Trial-1 (ctDNA+) Strata-1 (MSS/MMRp extendend RAS/RAFmut) Standard Therapy; Trial-1 (ctDNA+) Strata-1 (MSS/MMRp extendend RAS/RAFmut) Tailored Therapy; Trial-1 (ctDNA+) Strata-2 (MSI-H/MMRd & MSS/MMRp extended RAS/RAFwt) Standard Therapy; Trial-2 (ctDNA-) Standard Therapy
Drug: Folinic acid — Folinic acid is used as part of the FOLFOX chemotherapy regimen for patients with ctDNA+ results in the SAGITTARIUS trial. It is administered in the following way:
  FOLFOX Regimen: Folinic acid (leucovorin) 400 mg/m² is given intravenously on day 1, in combination with oxaliplatin 85 mg/m² IV on day 1 and fluorouracil 400 mg/m² IV bolus followed by 2400 mg/m² IV infusion over 46 hours, in each 14-day cycle.
  The dosage of folinic acid is standardized, while the duration of treatment can be adjusted based on patient response and liquid biopsy results, typically up to 6 months.
  Arms: Trial-1 (ctDNA+) Strata-1 (MSS/MMRp extendend RAS/RAFmut) Standard Therapy; Trial-1 (ctDNA+) Strata-1 (MSS/MMRp extendend RAS/RAFmut) Tailored Therapy; Trial-1 (ctDNA+) Strata-2 (MSI-H/MMRd & MSS/MMRp extended RAS/RAFwt) Standard Therapy; Trial-2 (ctDNA-) Standard Therapy
Drug: Fluorouracil — Fluorouracil is used as part of the FOLFOX chemotherapy regimen for patients with ctDNA+ results in the SAGITTARIUS trial. It is administered in the following way:
  FOLFOX Regimen: Fluorouracil 400 mg/m² is given as an intravenous (IV) bolus on day 1, followed by 2400 mg/m² as a continuous IV infusion over 46 hours, in combination with folinic acid (leucovorin) 400 mg/m² IV on day 1 and oxaliplatin 85 mg/m² IV on day 1. This regimen is repeated every 14 days.
  The dosage of fluorouracil is standardized, while the duration of treatment is typically up to 6 months, adjusted based on patient response and liquid biopsy results.
  Arms: Trial-1 (ctDNA+) Strata-1 (MSS/MMRp extendend RAS/RAFmut) Standard Therapy; Trial-1 (ctDNA+) Strata-1 (MSS/MMRp extendend RAS/RAFmut) Tailored Therapy; Trial-1 (ctDNA+) Strata-2 (MSI-H/MMRd & MSS/MMRp extended RAS/RAFwt) Standard Therapy; Trial-2 (ctDNA-) Standard Therapy
Drug: Temozolomide — Temozolomide is used as part of the tailored chemotherapy regimen for patients with ctDNA+ results in the SAGITTARIUS trial, specifically for those with MGMT-negative tumors. It is administered in the following way:
  TEMIRI Regimen: Temozolomide 150-200 mg/m² is taken orally once daily on days 1-5 of each 28-day cycle, in combination with irinotecan 250 mg/m² administered intravenously on day 1 of each cycle.
  The dosage of temozolomide is standardized, while the duration of treatment can be adjusted based on patient response and liquid biopsy results.
  Arms: Trial-1 (ctDNA+) Strata-1 (MSS/MMRp extendend RAS/RAFmut) Tailored Therapy
Drug: Irinotecan — Irinotecan is used as part of the tailored chemotherapy regimen for patients with ctDNA+ results in the SAGITTARIUS trial. It is administered in the following ways:
  TEMIRI Regimen: Irinotecan 250 mg/m² is administered intravenously on day 1 of each 28-day cycle, in combination with temozolomide 150-200 mg/m² taken orally once daily on days 1-5.
  FOLFIRI Regimen: Irinotecan 180 mg/m² is given intravenously on day 1, in combination with folinic acid (leucovorin) 400 mg/m² IV, fluorouracil 400 mg/m² IV bolus, followed by 2400 mg/m² IV infusion over 46 hours, in each 14-day cycle.
  The dosage of irinotecan is standardized, while the duration of treatment can be adjusted based on patient response and liquid biopsy results.
  Arms: Trial-1 (ctDNA+) Strata-1 (MSS/MMRp extendend RAS/RAFmut) Tailored Therapy
Drug: Nivolumab — Nivolumab is used as part of the tailored immunotherapy regimen for patients with ctDNA+ results, specifically for those with MSI-H/MMRd tumors in the SAGITTARIUS trial. It is administered in the following way:
  Nivolumab: 3 mg/kg is given intravenously every 2 weeks. This dosage is standardized, while the duration of treatment can be adjusted based on patient response and liquid biopsy results.
  Arms: Trial-1 (ctDNA+) Strata-2 (MSI-H/MMRd & MSS/MMRp extended RAS/RAFwt) Tailored Therapy
Drug: Ipilimumab — Ipilimumab is used as part of the tailored immunotherapy regimen for patients with ctDNA+ results, specifically for those with MSI-H/MMRd tumors in the SAGITTARIUS trial. It is administered in the following way:
  Ipilimumab: 1 mg/kg is given intravenously every 6 weeks. This dosage is standardized, while the duration of treatment can be adjusted based on patient response and liquid biopsy results.
  Arms: Trial-1 (ctDNA+) Strata-2 (MSI-H/MMRd & MSS/MMRp extended RAS/RAFwt) Tailored Therapy
Drug: Trastuzumab — Trastuzumab is used as part of the tailored targeted therapy regimen for patients with ctDNA+ results, specifically for those with HER2-amplified tumors in the SAGITTARIUS trial. It is administered in the following way:
  Trastuzumab: 8 mg/kg as an initial intravenous (IV) loading dose, followed by 6 mg/kg IV every 3 weeks.
  The dosage is standardized, while the duration of treatment can be adjusted based on patient response and liquid biopsy results.
  Arms: Trial-1 (ctDNA+) Strata-2 (MSI-H/MMRd & MSS/MMRp extended RAS/RAFwt) Tailored Therapy
Drug: Pertuzumab — Pertuzumab is used as part of the tailored targeted therapy regimen for patients with ctDNA+ results, specifically for those with HER2-amplified tumors in the SAGITTARIUS trial. It is administered in the following way:
  Pertuzumab: 840 mg as an initial intravenous (IV) loading dose, followed by 420 mg IV every 3 weeks.
  The dosage is standardized, while the duration of treatment can be adjusted based on patient response and liquid biopsy results.
  Arms: Trial-1 (ctDNA+) Strata-2 (MSI-H/MMRd & MSS/MMRp extended RAS/RAFwt) Tailored Therapy
Drug: Panitumumab — Panitumumab is used as part of the tailored targeted therapy regimen for patients with ctDNA+ results, specifically for those with multiple wild-type tumors (MSS/MMRp extended RAS/RAF wild-type) in the SAGITTARIUS trial. It is administered in the following way:
  Panitumumab: 6 mg/kg is given intravenously every 2 weeks. The dosage is standardized, while the duration of treatment can be adjusted based on patient response and liquid biopsy results.
  Arms: Trial-1 (ctDNA+) Strata-2 (MSI-H/MMRd & MSS/MMRp extended RAS/RAFwt) Tailored Therapy

SUMMARY:
Background & Rationale:

Colon cancer is a leading cause of cancer deaths, with a high recurrence rate in stage II high-risk and stage III patients due to undetectable micro-metastases. Liquid biopsy (LB) detects residual cancer DNA post-surgery and monitors treatment response.

Primary Objective:

Show that therapy based on tumor genetics and LB improves outcomes and quality of life for high-risk stage II and stage III colon cancer patients compared to conventional therapy.

Secondary Objectives:

Compare recurrence times. Evaluate side effects and quality of life. Assess cost differences. Validate LB accuracy.

Study Design: Patients are randomized into standard or personalized treatment groups based on LB results.

For positive LB results:

Randomized to standard or customized therapy. Monitor treatment response with LB.

For negative LB results:

Randomized to standard chemotherapy or follow-ups, starting treatment if a positive result appears.

Treatments:

Standard Chemotherapy:

CAPOX (capecitabine and oxaliplatin) FOLFOX (folinic acid, fluorouracil, and oxaliplatin)

Personalized Treatments:

Customized chemotherapy with CAPOX. Immunotherapy with nivolumab and ipilimumab. Targeted therapy with trastuzumab and pertuzumab. FOLFOX with anti-EGFR (epidermal growth factor receptor) therapy (panitumumab).

Population: 700 patients with operable stage III and high-risk stage II colon cancer.

Inclusion Criteria:

Aged 18 or older. Confirmed diagnosis. Tumor tissue sample available.

Exclusion Criteria:

History of other tumors within five years. Metastatic disease or recent experimental study participation. Major cardiovascular diseases, intestinal obstruction, autoimmune diseases, neuropathy, HIV (Human Immunodeficiency Virus), active TB (Tuberculosis), or hepatitis B/C infection.

Medical conditions contraindicating treatment. Prior neoadjuvant treatment administered before surgery.

Endpoints:

Primary:

Evaluate disease recurrence after two years.

Secondary:

Assess disease recurrence and overall survival at 3 and 5 years. Measure treatment safety and tolerability. Validate LB accuracy. Monitor quality of life using questionnaires.

The study will last 5 years and be conducted in 25-30 hospitals across Italy, Spain, and Germany.

DETAILED DESCRIPTION:
Background & Rationale:

Colon cancer (CC) is the second most lethal malignancy, accounting for nearly 10% of all cancer-related deaths. Despite over two-thirds of CC patients undergoing surgical resection, 50% of stage III patients relapse within 5 years. Adjuvant chemotherapy (ACT), typically involving oxaliplatin combined with a fluoropyrimidine, offers only a 10-15% survival advantage over 5-fluorouracil alone. The benefit from ACT is predicted by clinical and pathological parameters rather than metastatic propensity or biological sensitivity, and its success is limited by high toxicity levels, particularly oxaliplatin-induced peripheral sensory neuropathy.

Liquid biopsy (LB) profiling circulating tumor DNA (ctDNA) has emerged as an effective diagnostic tool for early cancer detection, staging, prognosis, monitoring drug resistance, and detecting minimal residual disease (MRD). Retrospective studies show that ctDNA detection post-surgery and post-ACT is associated with high recurrence risk and worse recurrence-free survival (RFS) in stage I-III colorectal cancer (CRC) patients. Prospective studies confirm ctDNA's prognostic value post-surgery and ACT.

SAGITTARIUS Trial Objectives:

Diagnosing MRD After Surgery: Utilize post-surgical LB to identify high-risk tumors and stratify stage II high-risk and stage III CC patients, enabling targeted treatments and reducing unnecessary chemotoxicity.

Establishing the Efficacy of Adjuvant Chemotherapy and Targeted Therapies: Tailor treatment based on the individual tumor genomic landscape to improve clinical outcomes and quality of life compared to conventional chemotherapy.

Study Design:

The SAGITTARIUS trial is a randomized phase III study designed to demonstrate the efficacy of ctDNA detection in guiding adjuvant clinical management of stage III and high-risk stage II CC patients. The trial employs the CE-IVD marked tumor-informed MRD assay Signatera (NATERA® Inc.) and comprehensive tumor genomic profiling (TruSight Oncology Comprehensive (EU), TSOComp, Illumina, Inc.). These tools will provide a detailed molecular genomic landscape of each patient's tumor, with results available within 8 weeks post-surgery for timely adjuvant treatment initiation.

Patient Stratification and Randomization:

Patients are stratified based on ctDNA status into two main trials:

Trial-1 (ctDNA Positive Patients): Includes further stratification based on MSS/MMRp extended RAS/RAF mutation status and MSI-H/MMRd status. Treatment arms include standard chemotherapy (CAPOX/FOLFOX) or personalized treatments with reassessment of ctDNA status guiding subsequent therapies.

Trial-2 (ctDNA Negative Patients): Patients are randomized to either a physician-choice chemotherapy regimen or intensive follow-up, with interventional LBs at specified intervals.

Therapeutic Approaches:

Standard Chemotherapy Regimens: CAPOX (capecitabine and oxaliplatin) and FOLFOX (folinic acid, fluorouracil, and oxaliplatin).

Personalized Therapies: Include options such as FOLFIRI or TEMIRI for RAS/RAF-mutated tumors, double immunotherapy (nivolumab and ipilimumab) for MSI-H/MMRd, anti-HER2 therapy (trastuzumab and pertuzumab) for HER2-amplified tumors, and FOLFOX combined with anti-EGFR (panitumumab) for multiple wild-type tumors.

Data Collection and Analysis:

Data will be collected through regular clinical evaluations, imaging studies, and questionnaires to assess various endpoints, including RFS, overall survival, treatment safety, tolerability, and quality of life. The primary endpoint is the 2-year RFS in ctDNA positive patients, while secondary endpoints include 3 and 5-year RFS, overall survival, and the accuracy of LB in detecting residual disease. Statistical analyses will follow the intention-to-treat principle, utilizing the Kaplan-Meier method for time-to-event data and stratified log-rank tests for comparison.

ELIGIBILITY:
Inclusion Criteria:

* SAGITTARIUS trial written informed consent.
* Age ≥ 18 years.
* Histologically confirmed diagnosis of operable stage III and High-Risk stage II CC located at least 12 cm from the anal verge by endoscopy and above the peritoneal reflection at surgery.
* Availability of the original FFPE tumor tissue.
* ECOG performance status 0-1.
* Normal organ functions (as defined in section 9.3).
* Women with childbearing potential (WOCBP) should complete a pregnancy test and be willing to use highly effective contraceptive methods.

Exclusion Criteria:

* History of another neoplastic disease, unless in remission for ≥ 5 years. Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (e.g., breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy are not excluded.
* Macroscopic or microscopic evidence of residual tumor (R1 or R2 resections). Patients should never have had any evidence of metastatic disease (including presence of tumor cells in the peritoneal lavage).
* Current or recent treatment with another investigational drug or participation in another investigational study.
* Patient unable to comply with the study protocol owing to psychological, social or geographical reasons.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the study.
* Inadequate contraception (male or female patients) if of childbearing or procreational potential.
* Clinically relevant cardiovascular disease.
* Acute or subacute intestinal occlusion or history of inflammatory bowel disease or any other autoimmune disease.
* Pre-existing neuropathy > grade 1. Known grade 3 or 4 allergic reaction to any of the components of the treatment.
* Has a known history of Human Immunodeficiency Virus (HIV).
* Has a known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus infection.
* Has a known history of active TB (Bacillus Tuberculosis).
* Has a medical condition that contraindicate the use of the investigational medicinal product (IMP) according to product indications.
* Prior neoadjuvant treatment administered before surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2024-10-22 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
2-Year Recurrence-Free Survival (RFS) | Assessed at 2 years post-surgery
  The primary outcome measure is the 2-year recurrence-free survival (RFS) rate, defined as the proportion of patients who remain free of disease recurrence two years after surgery. This metric is assessed using regular clinical evaluations and imaging studies. Recurrence is determined by the reappearance of colon cancer as confirmed by histological, radiological, or clinical findings.

SECONDARY OUTCOMES:
3-Year Recurrence-Free Survival (RFS) | Assessed at 3 years post-surgery
  The secondary outcome measure is the 3-year recurrence-free survival (RFS) rate, defined as the proportion of patients who remain free of disease recurrence three years after surgery. This metric is assessed using regular clinical evaluations and imaging studies. Recurrence is determined by the reappearance of colon cancer as confirmed by histological, radiological, or clinical findings.
5-Year Overall Survival (OS) | Assessed at 5 years post-surgery
  The secondary outcome measure is the 5-year overall survival (OS) rate, defined as the proportion of patients who are alive five years after surgery, regardless of disease status. This metric is assessed using regular clinical evaluations and follow-ups.
Treatment Safety and Tolerability | Assessed throughout the treatment period, up to 6 months
  This secondary outcome measure evaluates the safety and tolerability of the treatments, including both standard and personalized therapies. It involves recording and analyzing the incidence, severity, and type of adverse events experienced by patients during the treatment period, using the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Sensitivity and Specificity of Liquid Biopsy in Detecting Residual Disease | Assessed at regular intervals post-surgery, up to 2 years
  This outcome measure evaluates the effectiveness of liquid biopsy in detecting residual disease by comparing its results with traditional imaging techniques (CT scans, MRIs) and clinical findings. Sensitivity will be measured by the ability of liquid biopsy to correctly identify patients with residual disease, expressed as a percentage of positive results confirmed by imaging and clinical findings. Specificity will be measured by the ability to correctly identify patients without residual disease, also expressed as a percentage of negative results confirmed. The study will also assess the correlation between liquid biopsy results and traditional methods to ensure consistency in detecting residual disease.
Assessment of Quality of Life Using FACT-C Questionnaire | Assessed at regular intervals during the treatment period and during follow-up, up to 3 years or up to the date of first documented progression or the date of consent withdrawal
  This secondary outcome measure evaluates the impact of treatment on patients' quality of life specific to colorectal cancer using the Functional Assessment of Cancer Therapy-Colorectal (FACT-C) questionnaire. The FACT-C assesses quality of life across physical, social/family, emotional, and functional well-being domains. The questionnaire provides a score based on patient responses to various questions, with each question rated on a scale from 0 to 4, with higher scores indicating better quality of life.
Assessment of Quality of Life Using EQ-5D-5L Questionnaire | Assessed at regular intervals during the treatment period and during follow-up, up to 3 years or up to the date of first documented progression or the date of consent withdrawal
  This secondary outcome measure evaluates the impact of treatment on patients' quality of life across five dimensions using the EuroQol 5-Dimension 5-Level (EQ-5D-5L) questionnaire. The EQ-5D-5L evaluates quality of life in mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension is rated on a scale from 1 to 5, with 1 indicating no problems and 5 indicating extreme problems. The index score ranges from 0 to 1, with higher scores indicating better quality of life. Additionally, the EQ-5D-5L includes a visual analog scale (VAS) ranging from 0 (worst health imaginable) to 100 (best health imaginable) to assess the patient's overall health.

CONTACTS AND LOCATIONS:
Overall Officials: Clara Montagut, Principal Investigator — Hospital del Mar
Locations (26):
- Charité - Universitätsmedizin Berlin, Berlin, Germany
- Italy (12):
  - Azienda Sanitaria Locale di Biella, Biella, Biella
  - Fondazione Poliambulanza, Brescia, Brescia
  - Azienda Ospedaliera Universitaria San Martino, Genova, Genova
  - Istituto Europeo di Oncologia, Milan, Milano
  - Istituto Clinico Humanitas, Rozzano, Milano
  - Ospedale Niguarda, Milan, Milan
  - Ospedale Maggiore di Novara, Novara, Novara
  - Azienda Ospedaliera Universitaria di Parma, Parma, Parma
  - Ospedale Santa Maria della Misericordia, Perugia, Perugia
  - Azienda Unità Sanitaria Locale della Romagna, Ravenna, Ravenna
  - Policlinico Universitario Gemelli, Roma, Roma
  - Istituto di Candiolo, Candiolo, Torino
- Spain (13):
  - Hospital del Mar, Barcelona, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona, Barcelona
  - INCLIVA Instituto de Investigación Sanitaria, Valencia, Spain
  - Hospital Sant Pau Barcelona, Barcelona
  - Consorci Corporació Sanitària Parc Taulí, Barcelona
  - Instituto Catalán de Oncologia, Barcelona
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital Clinico Universitario San Carlos, Madrid
  - Complejo Hospitalario de Navarra, Pamplona
  - Hospital Universitario Marqués de Valdecilla, Santander
  - Hospital Clínico Universitario de Santiago, Santiago de Compostela
  - Hospital General Universitario de Valencia, Valencia
  - Hospital Universitario Miguel Servet, Zaragoza

IPD SHARING:
Plan to Share IPD: Undecided